CLINICAL TRIAL: NCT00930267
Title: Epidemiology and Etiology of Infections in Pediatric Cancer Patients: A Prospective Study
Brief Title: Infections in Pediatric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: yael12-HMO-CTIL
Record Dates: First submitted 2009-06-28; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Infections
Keywords: fever; children; cancer; leukemia; stem cell transplantation; infections in pediatric cancer patients presenting with fever during or following chemotherapy.
MeSH Terms: conditions — Infections; Fever; Neoplasms; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A prospective epidemiological study conducted in pediatric hematology oncology center in Hadassah medical center. The study will include all newly diagnosed pediatric cancer patients age 0-18 years admitted with fever during chemotherapy.

In each event of febrile episode during chemotherapy, the following data will be collected using a patient data form and computerized software.

Demographic data: age, gender, ethnicity. Clinical data: Underlying disease, immunizations, prophylactic antibiotics, presence of central venous catheter, intensity of chemotherapy, duration of fever, duration and severity of neutropenia, diagnosis of present event.

Imaging data Microbiological data Outcome The statistical analysis will be performed by an epidemiologist and statistician using the SPSS 12.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric cancer patients age 0-18 years admitted with fever during or following chemotherapy

Exclusion Criteria:

* No exclusions

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All newly diagnosed pediatric cancer patients age 0-18 years admitted with fever during or following chemotherapy
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Dan Engelhard, MD, Principal Investigator — Hadassah Medical Organization; Diana Averbuch, MD, Principal Investigator — Hadassah Medical Organization